CLINICAL TRIAL: NCT00068549
Title: A Phase I Study of Whole Pelvic Radiation Therapy With Concomitant Cisplatin and Gemcitabine Chemotherapy in Patients With Cervical Carcinoma (Stages I-IV) Limited to the Pelvis
Brief Title: Radiation Therapy Plus Cisplatin and Gemcitabine in Treating Patients With Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-9912; NCI-2012-02553 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000327715; GOG-9912 (Other: Gynecologic Oncology Group); GOG-9912 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Small Cell Carcinoma; Cervical Squamous Cell Carcinoma; Stage IB Cervical Cancer; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage IVA Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Gemcitabine; Cisplatin; Radiotherapy; Radiation; Brachytherapy

ARMS (1):
- Treatment (Experimental): Patients receive gemcitabine IV over 30 minutes and cisplatin IV over 1 hour on days 1, 8, 15, 22, 29, and 36 in the absence of disease progression or unacceptable toxicity. Patients also undergo external whole pelvis radiotherapy once daily on days 1-5, 8-13, 15-20, 22-27, and 29-34. After completion of external beam radiotherapy, patients undergo intracavitary radiotherapy and parametrial radiotherapy. The total elapsed time for completion of all radiotherapy is not more than 8 weeks.
  Interventions: Drug: Gemcitabine Hydrochloride; Drug: Cisplatin; Radiation: Radiation Therapy; Radiation: Internal Radiation Therapy

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdC; dFdCyd
Drug: Cisplatin — Given IV
Radiation: Radiation Therapy — Undergo whole pelvis radiotherapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RT
Radiation: Internal Radiation Therapy — Undergo brachytherapy
  Other Names: Brachytherapy; Internal Radiation; Internal Radiation Brachytherapy; Radiation Brachytherapy

SUMMARY:
This phase I trial is studying the side effects and best dose of gemcitabine when given together with radiation therapy and cisplatin in treating patients with cervical cancer that has not spread beyond the pelvis. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining cisplatin with gemcitabine may make the tumor cells more sensitive to radiation therapy and may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the toxicity of pelvic radiotherapy and concurrent cisplatin and gemcitabine in patients with cervical carcinoma limited to the pelvis.

II. Determine the maximum tolerated dose (MTD) of gemcitabine in combination with cisplatin and pelvic radiotherapy in these patients.

SECONDARY OBJECTIVES:

I. Determine the progression-free and overall survival of patients treated with gemcitabine at the MTD in this regimen.

II. Determine the site of recurrence, local versus distant, in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of gemcitabine.

Patients receive gemcitabine IV over 30 minutes and cisplatin IV over 1 hour on days 1, 8, 15, 22, 29, and 36 in the absence of disease progression or unacceptable toxicity. Patients also undergo external whole pelvis radiotherapy once daily on days 1-5, 8-13, 15-20, 22-27, and 29-34. After completion of external beam radiotherapy, patients undergo intracavitary radiotherapy and parametrial radiotherapy. The total elapsed time for completion of all radiotherapy is not more than 8 weeks.

Cohorts of 3-6 patients receive escalating doses of gemcitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 1 of 6 patients experiences dose-limiting toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary invasive carcinoma of the uterine cervix

  * Previously untreated disease
  * Any cell type
  * Stage IB_2, IIA, IIB, IIIA, IIIB, or IVA
* Para-aortic lymph nodes negative by radiologic evaluation or by biopsy if CT scan is suspicious for adenopathy
* No known metastases to scalene nodes or other organs outside the radiotherapy field
* Study enrollment within 8 weeks of diagnosis
* Performance status - GOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal
* Creatinine less than 2.0 mg/dL
* No renal abnormalities (e.g., pelvic kidney, horseshoe kidney, or renal transplantation) that would require modification of radiotherapy fields
* No ureteral obstruction allowed unless treated with stent or nephrostomy tube
* Not pregnant
* Fertile patients must use effective contraception
* No septicemia or severe infection
* No circumstance that would preclude study completion or follow-up
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No prior cytotoxic chemotherapy
* No prior pelvic or abdominal radiotherapy
* No prior therapy for this malignancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-10; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Incidence of acute toxicity using the 21 major categories of the CTEP CTC version 2.0 | Up to 30 days after completion of radiation therapy
Incidence of chronic toxicity using the CTC RTOG/EORTC late radiation morbidity scoring scheme | Up to 5 years
Dose of each drug | Up to 5 years
Number of cycles received | Up to 5 years

SECONDARY OUTCOMES:
Site (local/distant) of treatment failure | Up to 5 years
Progression-free survival | Up to 5 years
Overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rose, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States